CLINICAL TRIAL: NCT02727816
Title: Non-dispensing Fitting Study Comparing the Clinical Performance Hydrogel Sphere Design Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-65
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- filcon IV I (BC 8.6) / ocufilcon D (pair one) (Experimental): Participants were randomized to a test and control lens for each pair in a contralateral design.
  Interventions: Device: filcon IV I (BC 8.6); Device: ocufilcon D
- filcon IV I (BC 8.7) / ocufilcon D (pair two) (Experimental): Participants were randomized to a test and control lens for each pair in a contralateral design.
  Interventions: Device: filcon IV I (BC 8.7); Device: ocufilcon D
- methafilcon A (BC 8.6) / ocufilcon D (pair three) (Experimental): Participants were randomized to a test and control lens for each pair in a contralateral design.
  Interventions: Device: ocufilcon D; Device: methafilcon A (BC 8.6)
- methafilcon A (BC 8.7) / somofilcon A (pair four) (Experimental): Participants were randomized to a test and control lens for each pair in a contralateral design.
  Interventions: Device: methafilcon A (BC 8.7); Device: somofilcon A

INTERVENTIONS:
Device: filcon IV I (BC 8.6) — control lens
  Arms: filcon IV I (BC 8.6) / ocufilcon D (pair one)
Device: filcon IV I (BC 8.7) — control lens
  Arms: filcon IV I (BC 8.7) / ocufilcon D (pair two)
Device: ocufilcon D — test lens
  Arms: filcon IV I (BC 8.6) / ocufilcon D (pair one); filcon IV I (BC 8.7) / ocufilcon D (pair two); methafilcon A (BC 8.6) / ocufilcon D (pair three)
Device: methafilcon A (BC 8.6) — control lens
  Arms: methafilcon A (BC 8.6) / ocufilcon D (pair three)
Device: methafilcon A (BC 8.7) — control lens
  Arms: methafilcon A (BC 8.7) / somofilcon A (pair four)
Device: somofilcon A — test lens
  Arms: methafilcon A (BC 8.7) / somofilcon A (pair four)

SUMMARY:
The aim of this non-dispensing study is to evaluate the clinical performance of different hydrogel contact lens designs.

DETAILED DESCRIPTION:
This is a 35-subject, double masked, randomized, contra lateral, non-dispensing fitting trial comparing different hydrogel lens materials. For each study, this study will involve 2 visits: lens dispensing (baseline) and 1 hour post lens settling. Each subject will be randomized to wear the test and control lenses, in the right or left eye, in a series of four short fitting comparisons as follows:

Pair 1 (P1): filcon IV I (Base Curve (BC) 8.6) and ocufilcon D

Pair 2 (P2): filcon IV I (Base Curve (BC) 8.7) and ocufilcon D

Pair 3 (P3): methafilcon A (Base Curve (BC) 8.6) and ocufilcon D

Pair 4 (P4): methafilcon A (Base Curve (BC)8.7) and somofilcon A

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive).
* Has had a self-reported visual exam in the last two years.
* Is an adapted soft CL (Contact Lens) wearer.
* Has a CL spherical prescription between - 1.00 and - 6.00 (inclusive)
* Has a spectacle cylinder up to 0.75D (Diopters) in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease.
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule.
* Is willing to comply with the visit schedule.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a CL prescription outside the range of - 1.00 to - 6.00D
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities.
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GPC) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Participants were randomized to a test and control lens for each of the four lens pair in a contralateral design.
Period: Overall Study
Arm/Group | Overall Participants
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Centration - Pair One
Description: Centration for filcon IV I (Base Curve (BC) 8.6) / ocufilcon D (pair one) is assessed. (optimum, decentration acceptable, decentration unacceptable).
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of eyes
Groups:
- Filcon IV I (BC 8.6) - Pair One: Participants were randomized to a test and control lens for each pair in a contralateral design.
  filcon IV I (BC 8.6): control lens
- Ocufilcon D - Pair One: Participants were randomized to a test and control lens for each pair in a contralateral design.
  ocufilcon D: test lens
Arm/Group | Filcon IV I (BC 8.6) - Pair One | Ocufilcon D - Pair One
Number analyzed (Participants) | 35 | 35
number of eyes
  Baseline - Optimum | 35 | 35
  Baseline - Decentration acceptable | 0 | 0
  Baseline - Decentration unacceptable | 0 | 0
  1 hour - Optimum | 35 | 35
  1 hour - Decentration acceptable | 0 | 0
  1 hour - Decentration unacceptable | 0 | 0

2. Primary Outcome: Centration - Pair Two
Description: Centration for filcon IV I (Base Curve (BC) 8.7) / ocufilcon D (pair two) is assessed. (optimum, decentration acceptable, decentration unacceptable).
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of eyes
Groups:
- Filcon IV I (BC 8.7) - Pair Two: Participants were randomized to a test and control lens for each pair in a contralateral design.
  filcon IV I (BC 8.7): control lens
- Ocufilcon D - Pair Two: Participants were randomized to a test and control lens for each pair in a contralateral design.
  ocufilcon D: test lens
Arm/Group | Filcon IV I (BC 8.7) - Pair Two | Ocufilcon D - Pair Two
Number analyzed (Participants) | 35 | 35
number of eyes
  Baseline - Optimum | 35 | 35
  Baseline - Decentration acceptable | 0 | 0
  Baseline - Decentration unacceptable | 0 | 0
  1 hour - Optimum | 35 | 35
  1 hour - Decentration acceptable | 0 | 0
  1 hour - Decentration unacceptable | 0 | 0

3. Primary Outcome: Centration - Pair Three
Description: Centration for methafilcon A (Base Curve (BC) 8.6) / ocufilcon D (pair three) is assessed. (optimum, decentration acceptable, decentration unacceptable).
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of eyes
Groups:
- Filcon IV I (BC 8.6) - Pair Three: Participants were randomized to a test and control lens for each pair in a contralateral design.
  filcon IV I (BC 8.7): control lens
- Ocufilcon D - Pair Three: Participants were randomized to a test and control lens for each pair in a contralateral design.
  ocufilcon D: test lens
Arm/Group | Filcon IV I (BC 8.6) - Pair Three | Ocufilcon D - Pair Three
Number analyzed (Participants) | 35 | 35
number of eyes
  Baseline - Optimum | 35 | 35
  Baseline - Decentration acceptable | 0 | 0
  Baseline - Decentration unacceptable | 0 | 0
  1 hour - Optimum | 35 | 35
  1 hour - Decentration acceptable | 0 | 0
  1 hour - Decentration unacceptable | 0 | 0

4. Primary Outcome: Centration - Pair Four
Description: Centration for methafilcon A (Base Curve (BC) 8.7) / somofilcon A (pair four) is assessed. (optimum, decentration acceptable, decentration unacceptable).
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of eyes
Groups:
- Filcon IV I (BC 8.7) - Pair Four: Participants were randomized to a test and control lens for each pair in a contralateral design.
  filcon IV I (BC 8.7): control lens
- Somofilcon A - Pair Four: Participants were randomized to a test and control lens for each pair in a contralateral design.
  somofilcon A: test lens
Arm/Group | Filcon IV I (BC 8.7) - Pair Four | Somofilcon A - Pair Four
Number analyzed (Participants) | 35 | 35
number of eyes
  Baseline - Optimum | 35 | 35
  Baseline - Decentration acceptable | 0 | 0
  Baseline - Decentration unacceptable | 0 | 0
  1 hour - Optimum | 35 | 35
  1 hour - Decentration acceptable | 0 | 0
  1 hour - Decentration unacceptable | 0 | 0

5. Primary Outcome: Post-blink Movement - Pair One
Description: Post-blink movement for filcon IV I (BC 8.6) / ocufilcon D (pair one) is assessed. (0-5 Likert scale, 0=Insufficient, unacceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.6) - Pair One | Ocufilcon D - Pair One
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 6 | 5
  Minimum | 13 | 2
  Optimum | 16 | 28
  Moderate | 0 | 0
  Excessive | 0 | 0

6. Primary Outcome: Post-blink Movement - Pair One
Description: as for outcome 5
Time Frame: 1 hour
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.6) - Pair One | Ocufilcon D - Pair One
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 2 | 0
  Minimum | 19 | 9
  Optimum | 14 | 26
  Moderate | 0 | 0
  Excessive | 0 | 0

7. Primary Outcome: Post-blink Movement - Pair Two
Description: Post-blink movement for filcon IV I (BC 8.7) / ocufilcon D (pair two) is assessed. (0-5 Likert scale, 0=Insufficient, unacceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.7) - Pair Two | Ocufilcon D - Pair Two
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 3 | 2
  Minimum | 7 | 16
  Optimum | 15 | 14
  Moderate | 10 | 3
  Excessive | 0 | 0

8. Primary Outcome: Post-blink Movement - Pair Two
Description: as for outcome 7
Time Frame: 1 hour
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.7) - Pair Two | Ocufilcon D - Pair Two
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 4 | 1
  Minimum | 5 | 13
  Optimum | 23 | 20
  Moderate | 3 | 1
  Excessive | 0 | 0

9. Primary Outcome: Post-blink Movement - Pair Three
Description: Post-blink movement for methafilcon A (BC 8.6) / ocufilcon D (pair three) is assessed. (0-5 Likert scale, 0=Insufficient, unacceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.6) - Pair Three | Ocufilcon D - Pair Three
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 1 | 0
  Minimum | 8 | 9
  Optimum | 26 | 23
  Moderate | 0 | 3
  Excessive | 0 | 0

10. Primary Outcome: Post-blink Movement - Pair Three
Description: as for outcome 9
Time Frame: 1 hour
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.6) - Pair Three | Ocufilcon D - Pair Three
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 0 | 0
  Minimum | 10 | 5
  Optimum | 24 | 28
  Moderate | 1 | 2
  Excessive | 0 | 0

11. Primary Outcome: Post-blink Movement - Pair Four
Description: Post-blink movement for methafilcon A (BC 8.7) / somofilcon A (pair four) is assessed. (0-5 Likert scale, 0=Insufficient, unacceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.7) - Pair Four | Somofilcon A - Pair Four
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 7 | 9
  Minimum | 7 | 11
  Optimum | 18 | 14
  Moderate | 3 | 1
  Excessive | 0 | 0

12. Primary Outcome: Post-blink Movement - Pair Four
Description: as for outcome 11
Time Frame: 1 hour
Measure: Number; unit: number of eyes
Arm/Group | Filcon IV I (BC 8.7) - Pair Four | Somofilcon A - Pair Four
Number analyzed (Participants) | 35 | 35
number of eyes
  Insufficient | 3 | 1
  Minimum | 7 | 10
  Optimum | 25 | 24
  Moderate | 0 | 0
  Excessive | 0 | 0

13. Primary Outcome: Lens Tightness - Pair One
Description: Lens tightness on push on test for filcon IV I (BC 8.6) / ocufilcon D (pair one) is assessed. (0% - 100%, 100%=No movement, 50%=Optimum 0%=Falls from cornea without lid support)
Time Frame: Baseline and 1 hour
Measure: Mean (Standard Deviation); unit: Percent lens tightness
Arm/Group | Filcon IV I (BC 8.6) - Pair One | Ocufilcon D - Pair One
Number analyzed (Participants) | 35 | 35
Percent lens tightness
  Baseline | 62.8 (16.2) | 57.1 (15.8)
  1 hour | 64.9 (15.9) | 57.1 (14.5)

14. Primary Outcome: Lens Tightness - Pair Two
Description: Lens tightness on push on test for filcon IV I (BC 8.7) / ocufilcon D (pair two) is assessed. (0% - 100%, 100%=No movement, 50%=Optimum 0%=Falls from cornea without lid support)
Time Frame: Baseline and 1 hour
Measure: Mean (Standard Deviation); unit: percent lens tightness
Arm/Group | Filcon IV I (BC 8.7) - Pair Two | Ocufilcon D - Pair Two
Number analyzed (Participants) | 35 | 35
percent lens tightness
  Baseline | 57.0 (17.1) | 52.3 (16.5)
  1 hour | 57.7 (14.8) | 56.6 (17.1)

15. Primary Outcome: Lens Tightness - Pair Three
Description: Lens tightness on push on test for methafilcon A (BC 8.6) / ocufilcon D (pair three) is assessed. (0% - 100%, 100%=No movement, 50%=Optimum 0%=Falls from cornea without lid support)
Time Frame: Baseline and 1 hour
Measure: Mean (Standard Deviation); unit: percent lens tightness
Arm/Group | Filcon IV I (BC 8.6) - Pair Three | Ocufilcon D - Pair Three
Number analyzed (Participants) | 35 | 35
percent lens tightness
  Baseline | 54.0 (7.80) | 54.3 (10.7)
  1 hour | 54.3 (8.50) | 51.2 (6.60)

16. Primary Outcome: Lens Tightness - Pair Four
Description: Lens tightness on push on test for methafilcon A (BC 8.7) / somofilcon A (pair four) is assessed. (0% - 100%, 100%=No movement, 50%=Optimum 0%=Falls from cornea without lid support)
Time Frame: Baseline and 1 hour
Measure: Mean (Standard Deviation); unit: percent lens tightness
Arm/Group | Filcon IV I (BC 8.7) - Pair Four | Somofilcon A - Pair Four
Number analyzed (Participants) | 35 | 35
percent lens tightness
  Baseline | 61.1 (20.3) | 66.7 (19.9)
  1 hour | 56.3 (12.4) | 56.6 (11.6)

17. Primary Outcome: Overall Fit Preference - Pair One
Description: Investigator's lens fit acceptance / acceptability for filcon IV I (BC 8.6) / ocufilcon D (pair one) is assessed. Three choices: filcon IV I (BC 8.6), ocufilcon D, or no preference.
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of subjects
Arm/Group | Prefer Filcon IV I (BC 8.6) - Pair One | Prefer Ocufilcon D - Pair One | No Preference
Number analyzed (Participants) | 35 | 35 | 35
number of subjects
  Baseline | 4 | 15 | 16
  1 hour | 3 | 17 | 15

18. Primary Outcome: Overall Fit Acceptance - Pair Two
Description: Investigator's lens fit acceptance / acceptability for filcon IV I (BC 8.7) / ocufilcon D (pair two) is assessed. Three choices: filcon IV I (BC 8.7), ocufilcon D, or no preference.
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of subjects
Arm/Group | Prefer Filcon IV I (BC 8.7) - Pair Two | Prefer Ocufilcon D - Pair Two | No Preference
Number analyzed (Participants) | 35 | 35 | 35
number of subjects
  Baseline | 13 | 9 | 13
  1 hour | 13 | 6 | 16

19. Primary Outcome: Overall Fit Acceptance - Pair Three
Description: Investigator's lens fit acceptance / acceptability for methafilcon A (BC 8.6) / ocufilcon D (pair three) is assessed. Three choices: methafilcon A (BC 8.6), ocufilcon D, or no preference.
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of subjects
Arm/Group | Prefer Methafilcon A (BC 8.6) - Pair Three | Prefer Ocufilcon D - Pair Three | No Preference
Number analyzed (Participants) | 35 | 35 | 35
number of subjects
  Baseline | 12 | 6 | 17
  1 hour | 6 | 10 | 19

20. Primary Outcome: Overall Fit Acceptance - Pair Four
Description: Investigator's lens fit acceptance / acceptability for methafilcon A (BC 8.7) / somofilcon A (pair four) is assessed. Three choices: methafilcon A (BC 8.7), somofilcon A, or no preference.
Time Frame: Baseline and 1 hour
Measure: Number; unit: number of subjects
Arm/Group | Prefer Methafilcon A (BC 8.7) - Pair Four | Prefer Somofilcon A - Pair Four | No Preference
Number analyzed (Participants) | 35 | 35 | 35
number of subjects
  Baseline | 9 | 5 | 21
  1 hour | 12 | 8 | 15

ADVERSE EVENTS:
Arm/Group | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other